CLINICAL TRIAL: NCT03804580
Title: First-line Treatment With Osimertinib in EGFR-mutated Non-small Cell Lung Cancer, Coupled to Extensive Translational Studies
Brief Title: First-line Treatment With Osimertinib in EGFR-mutated Non-small Cell Lung Cancer
Acronym: FIOL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK 2018/1028
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
Keywords: Targeted therapy; EGFR
MeSH Terms: conditions — Lung Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- osimertinib (Experimental): All patients recieve osimertinib
  Interventions: Drug: osimertinib

INTERVENTIONS:
Drug: osimertinib — Non-randomized trial, all patients receive therapy

SUMMARY:
Phase II, single-arm study to assess the safety and efficacy of osimertinib (80 mg, orally, once daily) as first-line therapy in patients with EGFR mutation-positive, locally advanced or metastatic non-small cell lung cancer (NSCLC) who have not previously treated with an epidermal growth factor tyrosine kinase inhibitor agent.

DETAILED DESCRIPTION:
This is a phase II, single-arm study to assess the safety and efficacy of osimertinib (80 mg, orally, once daily) as first-line therapy in patients with EGFR mutation-positive, locally advanced or metastatic non-small cell lung cancer (NSCLC) who have not previously treated with an epidermal growth factor tyrosine kinase inhibitor agent.

Subjects will have to provide a biopsy sample (fresh or archival) for molecular testing at inclusion. If feasible, a biopsy will also be sampled when partial response is achieved and at the time of disease progression on osimertinib. Liquid biopsies will be sampled throughout the treatment period.

Subjects should continue on study treatment until RECIST 1.1-defined progression or until a treatment criterion is met. There is no maximum duration of treatment as subjects may continue to receive investigational product beyond RECIST1.1-defined progression as long as they are continuing to show clinical benefit, as judged by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent.
2. Age > 18 years.
3. Histologically or cytologically documented locally advanced or metastatic NSCLC not amenable to curative surgery or radiotherapy. Patients that have received systemic adjuvant therapy for non-metastatic disease in the past will need a new biopsy before inclusion.
4. Documented EGFR mutation in exon 18-21, except insertions in exon 20, based on tissue analysis.
5. ECOG status 0-2 and a minimum life expectancy of 12 weeks.
6. Patients with untreated, mild or moderately symptomatic and measurable brain metastases are eligible, but will be allocated to cohort A (see excl. point 6). Patients with pre-treated, stable and asymptomatic brain metastases will be allocated to cohort B.
7. At least one lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline according to RECIST 1.1.
8. Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women under 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with Luteinizing Hormone (LH) and Follicle-Stimulating Hormone (FSH) levels in the post-menopausal range for the institution
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
9. Male subjects must be willing to use barrier contraception.

Exclusion Criteria:

1. Previous systemic treatment against metastatic NSCLC.
2. Major surgery within 4 weeks of inclusion
3. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of inclusion
4. Subjects currently receiving (or unable to stop using) potent inducers of CYP3A4. Patients must stop using CYP3A4 inducers at least 3 weeks prior to treatment with osimertinib (see appendix A).
5. Subjects with spinal cord compression unless they have completed definitive therapy, are not on steroids and have had a stable neurological status for at least 2 weeks after completion of definitive therapy and steroids.
6. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
7. Previous malignancy (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, oesophageal, colon, endometrial, cervical, melanoma or breast) unless a complete remission was achieved at least 2 years prior to study entry.
8. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
9. Exclude based on any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
10. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
11. Inadequate bone marrow reserve or organ function (as demonstrated by any of the following laboratory values:

    * Absolute neutrophil count < 1.5 x 109/L
    * Platelet count < 100 x 109/L
    * Haemoglobin < 90 g/L
    * Alanine aminotransferase (ALT) > 2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases
    * Aspartate aminotransferase (AST) > 2.5 times ULN if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases
    * Total bilirubin > 1.5 times ULN if no liver metastases or > 3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases
    * Serum creatinine >1.5 times ULN concurrent with creatinine clearance <50 mL/min [measured or calculated by Cockcroft and Gault equation]-confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN
12. History of hypersensitivity of active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib.
13. Treatment with an investigational drug within five half-lives of the compound or 3 months, whichever is greater.
14. Previous enrolment in the present study or previous treatment with osimertinib.
15. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment, with the exception of alopecia and grade 2, prior platinum-therapy-related neuropathy.
16. Women who are pregnant or breast-feeding, or have a positive (urine or serum) pregnancy test prior to study entry
17. Involvement in the planning and/or conduct of the study (investigator staff and/or staff at the study site).
18. Judgment by the investigator that the subject should not participate in the study if the subject is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 12 weeks
  Measured by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Odd Terje Brustugun, MD PhD, Principal Investigator — Drammen Hospital - Vestre Viken
Locations (10):
- Denmark (4):
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- National Cancer Institute, Vilnius, Lithuania
- Norway (3):
  - Drammen Hospital - Vestre Viken HF, Drammen
  - Oslo University Hospital - Ullevaal, Oslo
  - St Olavs Hospital, Trondheim
- Sweden (2):
  - Lund University Hospital, Lund
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided